CLINICAL TRIAL: NCT00390676
Title: A Phase 1, Multicenter, Dose-Escalation Study to Investigate the Safety and Tolerability of ADH-1 in Combination With 1) Carboplatin or 2) Docetaxel or 3) Capecitabine in Subjects With N-Cadherin Positive, Advanced Solid Tumors (Adherex Protocol Number AHX-01-006)
Brief Title: A Study of ADH 1 in Combination With Carboplatin, or Docetaxel or Capecitabine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adherex Technologies, Inc. (Industry)
Collaborators: US Oncology Research (Industry)
Responsible Party: Clinical Study Manager, Adherex Technologies
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHX-01-006
Record Dates: First submitted 2006-10-18; First posted 2006-10-20 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Neoplasms
Keywords: cancer; tumors; anticarcinogenic agents; antineoplastic agents; cadherins; solid tumors
MeSH Terms: conditions — Neoplasms | interventions — Carboplatin; Docetaxel; Capecitabine

INTERVENTIONS:
Drug: ADH -1 and carboplatin
Drug: ADH -1 and docetaxel
Drug: ADH -1 and capecitabine

SUMMARY:
N-cadherin, a protein involved in blood vessel cell binding, is increased as cancer progresses, and is on the surface of many tumor cells. ADH-1 blocks N-cadherin. This study will test the safety and effects of the combination ADH-1 and carboplatin or ADH-1 and docetaxel or ADH-1 and capecitabine in subjects with specific incurable, solid tumors with a protein biomarker called N-cadherin.

ELIGIBILITY:
Inclusion criteria:

* Signed written informed consent
* Male and female patients > or = 18 years of age with a solid tumor(s) that is locally advanced or metastatic for which single agent carboplatin, or docetaxel or capecitabine would be appropriate
* Measurable disease
* Immunohistochemical evidence of N-cadherin expression in tumor tissue
* Adequate performance status and organ function, as evidenced by hematological and biochemical blood testing and ECG

Exclusion criteria:

* Receipt of ADH-1 prior to this clinical study
* Chemotherapy, radiotherapy, or any other investigational drug within 4 weeks before study entry
* History of spinal cord compression, or history of primary brain tumor(s) or brain metastases (known or suspected) unless any lesions have completely resolved following appropriate treatment and there has been no recurrence for at least 6 months
* History of tumors that have shown clinically significant evidence of active bleeding within 12 weeks before study entry
* Stroke, major surgery, or other major tissue injury within 4 weeks before study entry
* Uncontrolled congestive heart failure, coronary artery disease, or life threatening arrhythmias; myocardial infarction within 12 months; significant electrocardiogram (ECG) abnormalities, or known hypercoagulable states

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-11; Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Cancer Centers of Florida, Ocoee, Florida
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - New York Oncology Hematology P.C., Albany, New York
  - Dayton Oncology & Hematology, P.A, Kettering, Ohio
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Texas Oncology, PA, Dallas, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Cancer Specialists - Vancouver Cancer Center, Vancouver, Washington

REFERENCES:
- See also: Adherex Technologies Inc. Corporate Homepage — http://www.adherex.com